CLINICAL TRIAL: NCT05524259
Title: MYPP-trial: Myo-inositol Supplementation to Prevent Pregnancy Complications in Women With Polycystic Ovary Syndrome: a Multicentre Double-blind Randomised Controlled Trial
Brief Title: MYPP-trial: Myo-inositol Supplementation to Prevent Pregnancy Complications in Women With Polycystic Ovary Syndrome.
Acronym: MYPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, B.B. van Rijn, Associate Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MEC-2019-0005, NL67329.078.18
Record Dates: First submitted 2022-07-27; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes Mellitus; Preeclampsia; Preterm Birth; Polycystic Ovary Syndrome
MeSH Terms: conditions — Diabetes, Gestational; Pre-Eclampsia; Premature Birth; Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo-inositol and routinely recommended folic acid (Active Comparator): Myo-inositol is a naturally occurring substance, with a structure quite similar to glucose, which forms an essential component of the cell membrane and is known to support several cellular processes in all living organisms. It is present in nature in high abundance and can be found in many food products. Myo-inositol was historically considered part of the vitamin-B complex and can safely be used as a dietary supplement. In humans, it is synthesized de novo from glucose-6-phosphate in many tissues, mainly in the kidney. Under normal circumstances, the kidneys produce large quantities of myo-inositol, estimated at about 4 grams of endogenous production per day. Myo-inositol has been shown to have a physiological role in supporting the effects of insulin in all living beings. It fulfils a second messenger role in the insulin signalling pathway by enhancing the translocation of GLUT-4 receptors on the plasma membrane and thereby facilitates the intra-cellular uptake of glucose.
  Interventions: Dietary Supplement: Myo-inositol and routinely recommended folic acid
- Routinely recommended folic acid (Placebo Comparator): Folic acid supplements are part of routine pregnancy care and frequently used as background supplements in previous trials on myo-inositol supplementation in pregnancy.
  Interventions: Dietary Supplement: Routinely recommended folic acid

INTERVENTIONS:
Dietary Supplement: Myo-inositol and routinely recommended folic acid — Participants randomly allocated to the intervention group will receive 4 grams myo-inositol added to their routinely recommended 0.4 mg folic acid supplement, divided over two daily sachets of sugary powder throughout pregnancy.
  Arms: Myo-inositol and routinely recommended folic acid
Dietary Supplement: Routinely recommended folic acid — The control group will receive similar looking sachets of supplements containing only the standard dose of 0.4 mg folic acid without the added myo-inositol supplement as part of the current standard-of-care recommendation.
  Arms: Routinely recommended folic acid

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is the most common endocrine disorder in women of reproductive age. PCOS is a heterogeneous condition, characterised by metabolic disturbances, insulin resistance and hyperandrogenism. Pregnancies in women with PCOS have an increased risk of gestational diabetes mellitus, preeclampsia and preterm birth, and their offspring have an increased risk of aberrant birth weight and hospitalization. After pregnancy, PCOS is thought to have an impact on breastfeeding success and breastmilk composition.

Current strategies to improve pregnancy outcome among women with PCOS have not demonstrated significant risk reduction. Myo-inositol is a commonly used dietary supplement with a favourable effect on glucose metabolism and insulin sensitivity. Optimal intake of myo-inositol is associated with a decrease in glucose, lower insulin and lower testosterone levels in women with PCOS. Among women with PCOS-related disorders (e.g. in women with obesity), myo-inositol supplementation in pregnancy has been shown to have clinical benefits in preventing adverse pregnancy outcomes in a number of clinical trials, by reducing the risk of gestational diabetes mellitus, hypertensive complications and preterm birth.

The MYPP-trial will be the first randomised prospective trial aimed specifically at pregnant women with PCOS, to evaluate the potential effectiveness of myo-inositol supplementation as a nutritional intervention to prevent all three pregnancy complications associated with PCOS (i.e. GDM, preeclampsia and preterm birth). Secondary objectives are to evaluate the impact of supplementation on maternal (mental) and neonatal health, breastfeeding practices and breastmilk composition. In addition, a full cost-effectiveness analysis will be performed.

Women with a diagnosis of PCOS and a singleton pregnancy between 8+0 and 16+0 weeks of gestational age are eligible. Participants randomly allocated to the intervention group will receive 4 grams myo-inositol added to their routinely recommended folic acid supplement, divided over two daily sachets of sugary powder throughout pregnancy. The control group will receive similar looking sachets of supplements containing only the standard dose of folic acid without the added myo-inositol supplement, as part of the current standard-of-care recommendation. In addition to receiving supplements, participants will be asked to complete three questionnaires, provide blood and urine samples once each trimester of pregnancy, and routine ultrasound scanning will be performed to assess fetal growth. All study visits will be aligned with routine antenatal care appointments. Additionally, subjects can choose to participate in research on the impact of myo-inositol supplementation on breastfeeding and take part in the MYPP biobank.

The results of this study will provide important novel recommendations for PCOS patients on the importance of optimising life-style and nutrient intake to improve pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of PCOS according to the Rotterdam consensus criteria and confirmed by a gynaecologist
* A viable singleton pregnancy confirmed by ultrasound
* Being able to initiate the use of study supplements between 8+0 and 16+0 weeks gestational age
* Ability to understand Dutch or English
* Ability to provide written informed consent

Exclusion Criteria:

* Diagnosis of pre-existent type-1 or 2 diabetes mellitus
* Pre-existent renal failure, defined as an estimated glomerular filtration rate (eGFR) less than 50 ml/min/1.73m2
* Use of myo-inositol supplements, other insulin-mimetics, hypoglycaemic agents (e.g. metformin) and/or systemic steroids, that cannot be discontinued at the time of inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of PCOS patients in the two study arms that develop Gestational Diabetes Mellitus (GMD). | Measured from 12 weeks up to 28 weeks gestational age using an Oral Glucose Tolerance Test (OGTT)
  GDM is defined as any degree of glucose intolerance with onset or first recognition during pregnancy.
The incidence of PCOS patients in the two study arms that develop preeclampsia. | Measured from 20 weeks gestational age up to one week post-partum.
  Preeclampsia as defined by the International Society for the Study of Hypertension in Pregnancy (ISSHP).
The incidence of PCOS patients in the two study arm that give birth before 37 completed weeks of gestational age. | At delivery
  Preterm birth is internationally defined as any birth before 37 completed weeks of gestational age.

SECONDARY OUTCOMES:
Maternal mental health assessed by Beck Depression Inventory (BDI) Scale II Netherlands. | Measured at study inclusion, 36 weeks of pregnancy and 6 weeks postpartum.
  The BDI-II-NL measures characteristic attitudes and symptoms of depression and contains 21 items, subdivided in cognitive, affective and somatic factors. Patients rate themselves on these depressive symptoms by endorsing the most relevant statement (ranging in four steps of intensity from minimal to severe) covering a time frame of the past 2 weeks.
Maternal Health Related Quality of Life assessed by 5-Level EuroQol - five dimension (EQ-5D-5L) and Polycystic Ovary Syndrome Health-Related Quality of Life Questionnaire (PCOSQ) | Measured at study inclusion, 36 weeks of pregnancy and 6 weeks postpartum.
  he EQ-5D-5L records the patient's self-rated health, and a descriptive system. The descriptive system distinguishes five health domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The PCOSQ is the only existing validated, disease-specific, health related quality of life assessment questionnaire. As stated in the new evidence-based PCOS guidelines, this questionnaire could be clinically useful to highlight PCOS features causing greatest distress and was developed to evaluate the effect of treatment in clinical trials in PCOS.
The incidence of neonatal outcomes in the two study arms (e.g. incidence of neonatal intensive care unit (NICU) admissions, incidence of Neonatal hypoglycaemia). | Measured form birth and ultimately scored up until six weeks postpartum.
  * The incidence of Small-for-gestational-age (SGA): babies in the two study arms; birth weight ≤10th percentile or two standard deviations below the mean birth weight for gestational age, using Dutch Perinatal Registry birth weight reference charts.
  * The incidence of Large-for-gestational-age (LGA) babies in the two study arms: birth weight ≥90th percentile for gestational age, using Dutch Perinatal Registry birth weight reference charts.
  * The incidence of NICU admission in the two study arms, including reason for admission and time to discharge or transfer to another unit.
  * The incidence of Neonatal hypoglycaemia in the two study arms:

OTHER OUTCOMES:
Cost-effectiveness of myo-inositol supplementation using Health Technology Assessment (HTA) analyses. | Measured from study inclusion up until 6 weeks postpartum.
  To evaluate the cost-effectiveness of the nutritional intervention from a societal perspective, all resources used in maternity and neonatal care are recorded using questions derived from the Medical Consumption Questionnaire (MCQ).
Cost-effectiveness of myo-inositol supplementation using Health Technology Assessment (HTA) analyses. | Measured from study inclusion up until 6 weeks postpartum.
  To evaluate the patient perspective, questions derived from the EQ-5D-5L and the Productivity Cost Questionnaire (PCQ) are incorporated in the study questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://mypp-trial.nl/